CLINICAL TRIAL: NCT00928018
Title: A Phase III Multicenter, Randomized Trial Comparing Tacrolimus/Sirolimus/Methotrexate Versus Tacrolimus/Methotrexate or Cyclosporine/Mycophenolate Mofetil for GVHD Prophylaxis After Reduced Intensity Allogeneic Stem Cell Transplantation for Patients With Lymphoma
Brief Title: Tacrolimus/Sirolimus/Methotrexate vs Tacrolimus/Methotrexate or Cyclosporine/Mycophenolate Mofetil for GVHD Prophylaxis After Reduced Intensity Allogeneic Stem Cell Transplantation for Patients With Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Philippe Armand, MD, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-073; CA142106 (Other Grant/Funding Number: National Cancer Institute/NIH/DHHS)
Record Dates: First submitted 2009-06-24; First posted 2009-06-25 (Estimated); Results first posted 2015-12-18 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Non-hodgkin Lymphoma; Hodgkin Lymphoma
Keywords: allogeneic stem cell transplant; reduced intensity conditioning; graft versus host disease; GVHD; RIC transplantation
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Hodgkin Disease; Graft vs Host Disease | interventions — Sirolimus; Methotrexate; Tacrolimus; Cyclosporine; Cyclosporins; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sirolimus-Containing Regimen (Active Comparator): The Sirolimus containing arm will consist of the following drugs:
  Experimental Arm: tacrolimus + sirolimus + low-dose methotrexate
  Tacrolimus: Administered orally at a dose of 0.05 mg/kg based on ABW bid starting on day -3.
  Sirolimus:Given as a loading oral dose of 12 mg on day -3, then as a daily maintenance dose of 4 mg starting on day -2.
  Methotrexate: Administered by intravenous bolus infusion, per institutional standard, at a dose of 5 mg/m2 on days +1, +3 and +6.
  Interventions: Drug: Sirolimus; Drug: Methotrexate; Drug: Tacrolimus
- Sirolimus-Free regimen (Active Comparator): There are two choices for the Sirolimus free arm:
  Control Arm 1: tacrolimus + methotrexate
  Tacrolimus:Administered orally at a dose of 0.05 mg/kg based on ABW bid starting on day -3.
  Methotrexate:Administered by intravenous bolus infusion at a dose of 5 mg/m2 on days +1, +3 and +6. For patients receiving stem cells from unrelated donors, an additional dose will be given on day +11.
  Control Arm 2: cyclosporine + MMF
  Cyclosporine: administered orally at a dose of 6 mg/kg based on ABW bid starting on day -3.
  MMF:administered at a dose of 3gm daily orally (or intravenously if the patient cannot tolerate oral administration) divided in 2 or 3 doses (bid or tid) depending on physician preference starting on day 3.
  Interventions: Drug: Methotrexate; Drug: Tacrolimus; Drug: Cyclosporine; Drug: MMF

INTERVENTIONS:
Drug: Sirolimus — Taken orally for at least 12 months
  Other Names: Rapamycin
  Arms: Sirolimus-Containing Regimen
Drug: Methotrexate — Given intravenously on the first, third and sixth day after transplant
  Other Names: Abbreviated MTX; Trade name:Trexall
Drug: Tacrolimus — Taken orally or given intravenously for at least 6 months
  Other Names: Prograf
Drug: Cyclosporine — Taken orally or given intravenously for at least 6 months
  Other Names: Brand names:; •Gengraf; •Neoral; •Sandimmune; •Sangcya
  Arms: Sirolimus-Free regimen
Drug: MMF — Taken orally for about 2 months
  Other Names: Mycophenolate mofetil (MMF); Brand Names:; CellCept; Myfortic
  Arms: Sirolimus-Free regimen

SUMMARY:
This trial is comparing whether using a drug called sirolimus for graft versus host disease (GVHD) prevention can decrease the chance of the participant's lymphoma relapsing after transplantation, compared to using a standard GVHD prevention regimen without sirolimus. Since mTOR inhibitors have anti-lymphoma activity, their use after transplantation may lead to a decreased risk of relapse and hence better transplantation outcome.

DETAILED DESCRIPTION:
* Because no one knows which of the study options is best, participants will be "randomized" into one of the two possible groups for GVHD prophylaxis: 1) a sirolimus-containing regimen (tacrolimus, sirolimus and methotrexate) or 2) a sirolimus-free regimen (tacrolimus and methotrexate or cyclosporine and mycophenolate mofetil).
* Participants will receive a reduced intensity conditioning regimen. This is done to prepare the body for transplantation. This will consist of a combination of drugs (either fludarabine and busulfan or fludarabine, cyclophosphamide and low-dose total body irradiation). The purpose of these drugs is to weaken the immune system and lower the chance of the body rejecting the donated stem cells.
* Participants will also receive the GVHD prophylaxis regimen that they have been randomized to. These drugs will lower the chance of rejecting the donor cells and lower the chance of developing GVHD.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be eligible if their primary indication for transplantation is among the following: Indolent B-cell non-Hodgkin lymphoma (NHL); Aggressive B-Cell NHL; T-cell NHL; or Hodgkin Lymphoma.
* Patients must have one of the following combinations of disease status and disease histology at the time of enrollment: 1) Patients may be transplanted as part of first-line therapy if they have one of the following histologies: CLL with adverse cytogenetics, MCL or, T-cell NHL. 2) Patients may be transplanted as part of treatment for relapsed or refractory disease without a prior autologous transplantation of they have one of the following histologies: Indolent NHL (including CLL/SLL), MCL or T-cell NHL. 3) Patients may be transplanted as part of treatment for disease that has relapsed or progressed after autologous transplantation if they have any of the histologies listed above. Patients may also be enrolled without a prior autologous transplantation if they have a contraindication to autologous transplantation, in the opinion of the treating clinician. 4) There is no minimal or maximal time interval from the patient's last anti-lymphoma therapy and the time of transplantation.
* 18-72 years of age
* Matched related or matched unrelated donor
* Donor willing to donate peripheral blood stem cells and meeting institutional criteria for stem cell donation. The donor must be medically eligible to donate stem cells according to individual transplant center criteria.

Exclusion Criteria:

* Patients with Burkitt lymphoma or DLBCL with a c-myc rearrangement
* Karnofsky performance status of less than 70% at the time of registration
* Prior allogeneic stem cell transplantation (note that prior autologous stem cell transplantation is allowed)
* Uncontrolled infection
* Serum creatinine 2.0mg/dl or greater
* Total bilirubin 2.0mg/dl or greater (unless related to hemolysis or Gilbert's syndrome)
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) 3 times or greater than the institutional upper limit of normal
* Left ventricular ejection fraction < 30%
* Cholesterol > 500mg/dl or triglycerides > 500 mg/dl despite appropriate treatment
* Seropositivity for HIV
* Pregnancy or breast-feeding (effective contraception must be used during therapy and for at least 6 months after the end of immunosuppressive agents)
* Prior history of allergy to sirolimus, tacrolimus, cyclosporine, methotrexate or MMF
* Concomitant treatment with another investigational drug (unless cleared by study chair)

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2009-06; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Armand, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (5):
- United States (5):
  - Emory University Hospital, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Ohio State University, Columbus, Ohio

REFERENCES:
- [Derived] Armand P, Kim HT, Sainvil MM, Lange PB, Giardino AA, Bachanova V, Devine SM, Waller EK, Jagirdar N, Herrera AF, Cutler C, Ho VT, Koreth J, Alyea EP, McAfee SL, Soiffer RJ, Chen YB, Antin JH. The addition of sirolimus to the graft-versus-host disease prophylaxis regimen in reduced intensity allogeneic stem cell transplantation for lymphoma: a multicentre randomized trial. Br J Haematol. 2016 Apr;173(1):96-104. doi: 10.1111/bjh.13931. Epub 2016 Jan 5. PMID 26729448

RESULTS

PARTICIPANT FLOW:
Groups:
- Sirolimus-Containing Regimen: The Sirolimus containing arm will consist of the following drugs:
  Experimental Arm: tacrolimus + sirolimus + low-dose methotrexate
  Tacrolimus: Administered orally at a dose of 0.05 mg/kg based on ABW bid starting on day -3.
  Sirolimus:Given as a loading oral dose of 12 mg on day -3, then as a daily maintenance dose of 4 mg starting on day -2.
  Methotrexate: Administered by intravenous bolus infusion, per institutional standard, at a dose of 5 mg/m2 on days +1, +3 and +6.
  Sirolimus: Taken orally for at least 12 months
  Methotrexate: Given intravenously on the first, third and sixth day after transplant
  Tacrolimus: Taken orally or given intravenously for at least 6 months
- Sirolimus-Free Regimen: There are two choices for the Sirolimus free arm:
  Control Arm 1: tacrolimus + methotrexate
  Tacrolimus:Administered orally at dose of 0.05 mg/kg based on ABW bid starting on day -3.
  Methotrexate:Administered by intravenous bolus infusion at dose of 5 mg/m2 on days +1, +3 and +6. For patients receiving stem cells from unrelated donors, an additional dose will be given on day +11.
  Control Arm 2: cyclosporine + MMF
  Cyclosporine: administered orally at dose of 6 mg/kg based on ABW bid starting on day -3.
  MMF:administered at dose of 3gm daily orally (or intravenously if the patient cannot tolerate oral administration) divided in 2 or 3 doses (bid or tid) depending on physician preference starting day 3.
  Methotrexate: Given intravenously on the first, third and sixth day after transplant
  Tacrolimus: Taken orally or given intravenously for at least 6 months
  Cyclosporine: Taken orally or given intravenously for at least 6 months
  MMF: Taken orally for about 2 months
Period: Overall Study
Arm/Group | Sirolimus-Containing Regimen | Sirolimus-Free Regimen
Started | 66 (One Arm A patient withdrew consent, treated as Arm B, but analyzed on Arm A based on intent-to-treat) | 73
Completed | 65 | 73
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sirolimus-Containing Regimen | Sirolimus-Free Regimen | Total
Number analyzed (Participants) | 66 | 73 | 139
Age, Continuous [Median (Full Range); unit: years] | 58 [23 to 70] | 57 [23 to 69] | 57 [23 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 29 | 53
  Male | 42 | 44 | 86
Region of Enrollment [Number; unit: participants]
  United States | 66 | 73 | 139

OUTCOME MEASURES:

1. Primary Outcome: To Compare 2-year Overall Survival of Patients With Lymphoma Undergoing RIC SCT Between Those Receiving Tacrolimus/Sirolimus/Methotrexate and Those Receiving Tacrolimus/Methotrexate or Cyclosporine/Mycophenolate Mofetil
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sirolimus-Containing Regimen | Sirolimus-Free Regimen
Number analyzed (Participants) | 66 | 73
percentage of participants | 70 [57 to 79] | 68 [57 to 78]

2. Secondary Outcome: To Compare 2-year Progression-free Survival Between the Two Treatment Arms
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sirolimus-Containing Regimen | Sirolimus-Free Regimen
Number analyzed (Participants) | 66 | 73
percentage of participants | 61 [48 to 71] | 58 [45 to 68]

3. Secondary Outcome: To Compare the 2-year Cumulative Incidences of Disease Progression and of Non-relapse Mortality Between the Two Treatment Arms
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sirolimus-Containing Regimen | Sirolimus-Free Regimen
Number analyzed (Participants) | 66 | 73
percentage of participants
  Cumulative incidence of relapse/progression | 26 [16 to 37] | 30 [20 to 41]
  Non-relapse mortality | 14 [7 to 23] | 12 [6 to 21]

4. Secondary Outcome: To Compare the 180-day Cumulative Incidence of Grades II-IV and Grades III-IV Acute GVHD Between the Two Treatment Arms
Time Frame: 6 months
Measure: Number; unit: percentage of participants
Arm/Group | Sirolimus-Containing Regimen | Sirolimus-Free Regimen
Number analyzed (Participants) | 66 | 73
percentage of participants
  Grade II-IV aGVHD | 9 | 25
  Grade III-IV aGVHD | 3 | 4

5. Secondary Outcome: To Compare the 2-year Cumulative Incidence of Chronic GVHD Between the Two Treatment Arms.
Time Frame: 2 years
Measure: Number; unit: percentage of participants
Arm/Group | Sirolimus-Containing Regimen | Sirolimus-Free Regimen
Number analyzed (Participants) | 66 | 73
percentage of participants | 59 | 63

6. Secondary Outcome: To Compare the 2-year of Overall Survival, Progression-free Survival, Cumulative Incidences of Progression and Non-relapse Mortality Between the Treatment Arms for Each Histology Studied.
Time Frame: 2 years
Population: Given the small number of patients within each group, we considered indolent histologies (indolent B-cell NHL, CLL and HL) together in one group (indolent group), and aggressive histologies (aggressive B-cell NHL, MCL, and T-cell NHL) in another (aggressive group).
Measure: Number; unit: percentage of participants
Groups:
- Indolent Group: Sirolimus-Containing Regimen: Indolent group:indolent B-cell NHL, CLL and HL histologies
  The Sirolimus containing arm will consist of the following drugs:
  Experimental Arm: tacrolimus + sirolimus + low-dose methotrexate
  Tacrolimus: Administered orally at a dose of 0.05 mg/kg based on ABW bid starting on day -3.Taken orally or given intravenously for at least 6 months
  Sirolimus:Given as a loading oral dose of 12 mg on day -3, then as a daily maintenance dose of 4 mg starting on day -2.Taken orally for at least 12 months
  Methotrexate: Administered by intravenous bolus infusion, per institutional standard, at a dose of 5 mg/m2 on days +1, +3 and +6.Given intravenously on the first, third and sixth day after transplant
- Indolent Group: Sirolimus-Free Regimen: Indolent group: indolent B-cell NHL, CLL and HL histologies
  There are two choices for the Sirolimus free arm:
  Control Arm 1: tacrolimus + methotrexate
  Tacrolimus:Administered orally at dose of 0.05 mg/kg based on ABW bid starting on day -3. Taken orally or given intravenously for at least 6 months
  Methotrexate:Administered by intravenous bolus infusion at dose of 5 mg/m2 on days +1, +3 and +6. For patients receiving stem cells from unrelated donors, an additional dose will be given on day +11.
  Control Arm 2: cyclosporine + MMF
  Cyclosporine: administered orally at dose of 6 mg/kg based on ABW bid starting on day -3. Taken orally or given intravenously for at least 6 months
  MMF:administered at dose of 3gm daily orally (or intravenously if the patient cannot tolerate oral administration) divided in 2 or 3 doses (bid or tid) depending on physician preference starting day 3. Taken orally for about 2 months.
- Aggressive Group: Sirolimus-Containing Regimen: Aggressive group: aggressive B-cell NHL, MCL, and T-cell NHL histologies
  The Sirolimus containing arm will consist of the following drugs:
  Experimental Arm: tacrolimus + sirolimus + low-dose methotrexate
  Tacrolimus: Administered orally at a dose of 0.05 mg/kg based on ABW bid starting on day -3.Taken orally or given intravenously for at least 6 months
  Sirolimus:Given as a loading oral dose of 12 mg on day -3, then as a daily maintenance dose of 4 mg starting on day -2.Taken orally for at least 12 months
  Methotrexate: Administered by intravenous bolus infusion, per institutional standard, at a dose of 5 mg/m2 on days +1, +3 and +6.Given intravenously on the first, third and sixth day after transplant
- Aggressive Group: Sirolimus-Free Regimen: Aggressive group: aggressive B-cell NHL, MCL, and T-cell NHL histologies
  There are two choices for the Sirolimus free arm:
  Control Arm 1: tacrolimus + methotrexate
  Tacrolimus:Administered orally at dose of 0.05 mg/kg based on ABW bid starting on day -3. Taken orally or given intravenously for at least 6 months
  Methotrexate:Administered by intravenous bolus infusion at dose of 5 mg/m2 on days +1, +3 and +6. For patients receiving stem cells from unrelated donors, an additional dose will be given on day +11.
  Control Arm 2: cyclosporine + MMF
  Cyclosporine: administered orally at dose of 6 mg/kg based on ABW bid starting on day -3. Taken orally or given intravenously for at least 6 months
  MMF:administered at dose of 3gm daily orally (or intravenously if the patient cannot tolerate oral administration) divided in 2 or 3 doses (bid or tid) depending on physician preference starting day 3. Taken orally for about 2 months.
Arm/Group | Indolent Group: Sirolimus-Containing Regimen | Indolent Group: Sirolimus-Free Regimen | Aggressive Group: Sirolimus-Containing Regimen | Aggressive Group: Sirolimus-Free Regimen
Number analyzed (Participants) | 38 | 40 | 28 | 33
percentage of participants
  Overall Survival | 82 | 63 | 54 | 76
  Progression Free Survival | 71 | 53 | 46 | 64
  Cumulative Incidence of Progression | 21 | 33 | 32 | 27
  Non-relapse mortality | 8 | 15 | 21 | 9

ADVERSE EVENTS:
Time Frame: Participating investigators will assess the occurrence of AEs and SAEs at all participant evaluation time points during the study. The study defined follow up period is 2 years.
Description: All AEs grades 3-5 and SAEs whether reported by participant, discovered during questioning, directly observed, or detected by physical examination, laboratory test, etc, will be recorded in participant's medical record and appropriate study-specific forms
  Only events reported in >1 patient on at least one of the arms are listed in Other AE table
Arm/Group | Sirolimus-Containing Regimen | Sirolimus-Free Regimen
Serious Adverse Events (participants affected / at risk) | 15/66 | 15/73
Other Adverse Events (participants affected / at risk) | 41/66 | 54/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sirolimus-Containing Regimen (N=66) | Sirolimus-Free Regimen (N=73)
Other: Relapse/Progressive disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
GVHD (Immune system disorders) | 0 (0) | 4 (4)
Treatment Related Secondary Malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombotic Microangiopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 0 (0) | 1 (1)
Heart Failure (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular and Nodal Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 1 (1)
Obstuction--GI, small bowel (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Edema (General disorders) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 0 (0) | 1 (1)
Liver failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Other- Systemic inflammatory response syndrome (SIRS) (Immune system disorders) | 0 (0) | 1 (1)
Leukopenia (Investigations) | 0 (0) | 1 (1)
Thrombocytopenia (Investigations) | 2 (2) | 0 (0)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Altered mental status (Nervous system disorders) | 0 (0) | 2 (2)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Hemorrhage, CNS (cerebrovascular) (Nervous system disorders) | 0 (0) | 1 (1)
Confusion (Nervous system disorders) | 0 (0) | 2 (2)
Acute Kidney Injury/Renal Failure (Renal and urinary disorders) | 3 (3) | 1 (1)
Adult Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Other--Respiratory failure/lung injury (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Other--Stroke (Vascular disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Vascular disorders) | 2 (2) | 2 (2)
Infection (Infections and infestations) | 8 (11) | 6 (6)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sirolimus-Containing Regimen (N=66) | Sirolimus-Free Regimen (N=73)
TMA/renal failure/hemolysis (Renal and urinary disorders) | 12 (12) | 6 (6)
Neutropenia (Blood and lymphatic system disorders) | 12 (12) | 16 (16)
Thrombocytopenia (Investigations) | 11 (11) | 14 (14)
Leukopenia (Investigations) | 6 (6) | 8 (8)
Infection (Infections and infestations) | 3 (3) | 17 (17)
Hyperlipidemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Anorexia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Cataract (Eye disorders) | 2 (2) | 1 (1)
Confusion/psychosis/encephalopathy (Nervous system disorders) | 8 (8) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 4 (4)
Hematoma (Vascular disorders) | 2 (2) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 10 (10)
Hepatic (Hepatobiliary disorders) | 4 (4) | 15 (15)
Stomatitis/mucositis (Gastrointestinal disorders) | 1 (1) | 4 (4)
Nausea/vomiting (Gastrointestinal disorders) | 4 (4) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 5 (5)
Neuropathy (Nervous system disorders) | 4 (4) | 0 (0)
Weakness (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1) | 8 (8)
Allergic Reaction (Immune system disorders) | 0 (0) | 2 (2)
Cardiac (Cardiac disorders) | 3 (3) | 7 (7)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Pain (Nervous system disorders) | 1 (1) | 8 (8)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypotension (Cardiac disorders) | 1 (1) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes